CLINICAL TRIAL: NCT05726591
Title: A Phase I/II Trial Evaluating Long-Term Use of a Pediatric Robotic Exoskeleton (P.REX/Agilik) to Improve Gait in Children With Movement Disorders
Brief Title: Evaluating Long-term Use of a Pediatric Robotic Exoskeleton (P.REX/Agilik) to Improve Gait in Children With Movement Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10001180; 001180-CC
Record Dates: First submitted 2023-02-11; First posted 2023-02-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10-23

CONDITIONS: Cerebral Palsy; Muscular Dystrophy; Spina Bifida; Incomplete Spinal Cord Injury
Keywords: EEG; Muscular Dystophies; Cerebral Palsy; Knee; incomplete spinal cord injury
MeSH Terms: conditions — Cerebral Palsy; Muscular Dystrophies; Spinal Dysraphism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 12 weeks-study intervention
  Interventions: Device: EA-KAFO
- Group B (No Intervention): 12 weeks the control first.

INTERVENTIONS:
Device: EA-KAFO — This study tests a single device that contains multiple potential configurations as outlined in Table 1 of the protocol. Each participant be evaluated in multiple configurations, minimally including the baseline configuration and the motor assist condition at the knee.
  Arms: Group A

SUMMARY:
Background:

People with cerebral palsy, spina bifida, muscular dystrophy, or spinal cord injury often have muscle weakness and problems controlling how their legs move. This can affect how they walk. The NIH has designed a robotic device (exoskeleton) that can be worn on the legs while walking. The wearable robot offers a new form of gait training.

Objective:

To learn whether a robotic device worn on the legs can improve walking ability in those with a gait disorder.

Eligibility:

People aged 3 to 17 years with a gait disorder involving the knee joint.

Design:

Participants will be screened. They will have a physical exam. Their walking ability will be tested.

Participants will have markers taped on their body; they will walk while cameras record their movements. They will undergo other tests of their motor function and muscle strength.

The study will be split into three 12-week phases. During 1 phase, participants will continue with their standard therapy.

During another phase, participants will work with the exoskeleton in a lab setting. Their legs will be scanned to create an exoskeleton with a customized fit. The exoskeleton operates in different modes: in exercise mode, it applies force that makes it difficult to take steps; in assistance mode, it applies force meant to aid walking; in combination mode, it alternates between these two approaches.

During the third phase, participants may take the exoskeleton home. They will walk in the device at least 1 hour per day, 5 days per week, for 12 weeks.

Participants walking ability will be retested after each phase....

DETAILED DESCRIPTION:
Study Description:

This randomized crossover trial will determine whether 12 weeks of overground gait training with a robotic exoskeleton outside of the clinical setting has a beneficial effect on walking ability, muscle activity, and overall gross motor function. Participants will be randomized into two groups, one that receives the exoskeleton therapy first before crossing over to continue standard therapy and one that continues standard therapy before completing the exoskeleton intervention. An in-lab training and accommodation period will be completed prior to the exoskeleton being sent home for use outside the clinical setting. We will monitor exoskeleton use during the intervention period for compliance and safety. Assessments of gait biomechanics, neuromuscular activity and functional mobility will be completed before and after the intervention and at 6 weeks post- intervention. It is hypothesized that the 12-week exoskeleton intervention outside the clinic setting will show greater improvements than the standard therapy.

Objectives:

Primary Objective: To evaluate the effectiveness of a longitudinal robotic exoskeleton gait training paradigm in improving crouch gait from CP or knee extension deficiency from SB, iSCI or MD in children, assessed as improvement in knee angle during walking before and after the intervention period.

Secondary Objectives:

To evaluate changes in muscle strength and gait speed following longitudinal intervention with robotic exoskeleton in children with crouch gait from CP or knee extension deficiency from SB, iSCI or MD. Additionally, to evaluate the primary endpoint of knee joint range of motion at multiple time points to assess for order effect and persistence of any observed effect.

Exploratory Objectives:

To assess the effect of exoskeleton dosage (i.e., time spent using the device) on the primary endpoint.

Additionally, to evaluate change in knee extensor and flexor muscle spasticity following longitudinal intervention with a robotic exoskeleton in children with crouch gait from CP or knee extension deficiency from SB, iSCI or MD. Additionally, to asses improvement in gross motor function following the same intervention. Finally, to evaluate the safety and feasibility of a community-based protocol for rehabilitation using a pediatric robotic exoskeleton.

Endpoints:

Primary Endpoint: Knee extension as assessed by peak knee angle during midstance phase of walking.

Secondary Endpoints: Change in knee extensor muscle activation and strength after exoskeleton intervention; Change in average gait speed after exoskeleton intervention; Persistence of the primary endpoint (change in knee angle) at 6 weeks post intervention; Effect of order of standard therapy and exoskeleton intervention.

Exploratory Endpoints:

Effect of exoskeleton intervention dosage on change in peak knee angle during walking; Change in knee extensor and flexor spasticity after exoskeleton intervention; Improvement in gross motor function after exoskeleton intervention; Feasibility and safety of exoskeleton use outside clinical setting assessed by participant compliance and occurrence of adverse events, respectively.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated separate informed consent and assent forms for screening purposes. Upon inclusion in the protocol, provision of signed and dated informed consent and assent forms to begin participation in the study will be necessary.
* Stated willingness to comply with all study procedures and availability for the duration of the study, or alternatively, ability to do so based on parent report and physician observation during history and physical examination.
* Age 3 to 17 years old.
* Have a gait pathology involving the knee joint, from a diagnosis of cerebral palsy, muscular dystrophy, spina bifida, or incomplete spinal cord injury.
* Knee joint range of motion of at least 25 degrees in the sagittal plane (knee extension/flexion) assessed with hip extended in supine position. Hamstring contracture as assessed by straight leg raising test does not limit ability to participate in the study.
* Ankle joint range of motion of at least 15 degrees in the sagittal plane (dorsi-plantar flexion) with the foot in neutral alignment.
* A measured foot-thigh angle of -15 to 30 degrees in prone position.
* Able to walk at least 10 feet without stopping with or without a walking aid.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Any neurological, musculoskeletal or cardiorespiratory injury, health condition, or diagnosis other than cerebral palsy, muscular dystrophy, spina bifida, or incomplete spinal cord injury that would affect the ability to walk as directed with the robotic exoskeleton.
* A history of uncontrolled seizure in the past year.
* Pregnancy. A urine test will be performed for all participants who are able to become pregnant at the initial screening visit and in the case of a positive test, the participant will be excluded from participation. Further monitoring will rely on self-reporting of interruption in menstruation that would require re-testing for pregnancy at the next visit.
* Any acute cardiopulmonary condition which limits exercise to less than 60 minutes per session or less than 5 days per week.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of a longitudinal exoskeleton training program in the community, as opposed to a standard regimen of therapy of the same magnitude, at improving knee extension deficiency in children with CP, SB, iSCI or MD. | 36 Weeks
  The primary endpoint will be knee extension range of motion. This will be assessed using knee angle at two positions in the gait cycle: knee angle at initial contact and peak knee angle during stance

SECONDARY OUTCOMES:
To evaluate improvement in overground walking of children with CP, SB, iSCI or MD as a function of average gait speed while walking with the robotic exoskeleton | 15 Weeks
  This outcome will be measured using peak and mean activation of knee extensor and knee flexor muscles during walking.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Bulea, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Derived] Devine TM, Alter KE, Damiano DL, Bulea TC. A randomized cross-over study protocol to evaluate long-term gait training with a pediatric robotic exoskeleton outside the clinical setting in children with movement disorders. PLoS One. 2024 Jul 8;19(7):e0304087. doi: 10.1371/journal.pone.0304087. eCollection 2024. PMID 38976710
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001180-CC.html